CLINICAL TRIAL: NCT01365546
Title: Prospective, Open-Label, Multi-Center, Phase III CLinical Study to Investigate the Efficacy and Safety of Human Factor VWF/FVIII Concentrate (Wilate) in Subjects With Inherited Von Willebrand Disease Who Undergo Surgical Procedures
Brief Title: Wilate in Subjects With Von Willebrand Disease Who Undergo Surgery
Acronym: WONDERS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Wil-24
Record Dates: First submitted 2011-05-27; First posted 2011-06-03 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Prevent Bleeding in Major Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- human VWF/FVIII concentrate (Experimental)
  Interventions: Biological: human VWF/FVIII concentrate

INTERVENTIONS:
Biological: human VWF/FVIII concentrate — intravenous infusion. Dose based on subject's individual invivo-recovery

SUMMARY:
Proportion of surgeries in which the primary endpoint (overall assessment) is classified as success.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with congenital VWD (von Willebrand Disease)
* Require therapy with a VWF (von Willebrand Factor) product to treat any major surgical procedure

Exclusion Criteria:

* Known coagulation disorder other than VWD
* Known history of, or suspected VWF or FVIII inhibitors
* Subjects with hepatic liver disease
* Known or suspected hypersensitivity or previous evidence of severe side effects to wilate or other VWF/FVIII concentrates
* Pregnant women in the first 20 weeks of gestation

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (3):
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - UNC-CH Comprehensive Hemophilia Center, Chapel Hill, North Carolina
  - Blood Center of Wisconsin, Milwaukee, Wisconsin
- SHAT Joan Pavel, Sofia, Bulgaria
- India (2):
  - Sahyadri Specialty Hospital, Pune, Pune
  - Christian Medical College, Vellore, Tamil Nadu
- Italy (3):
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Granda Ospedale Maggiore Policlinico, Milan
  - ULSS6 Vicenza Ematologia, Vicenza
- Sultan Quaboos University Hospital, Muscat, Oman
- Instytut Hematologii i Transfuzjologii, Warsaw, Poland
- Romania (2):
  - Fundeni Clinical Institute, Bucharest
  - Louis Turcanu Childrens Emergency Hospital, Timișoara
- Hemophilia Comprehensive Care Center, Johannesburg, South Africa
- Ege University, Izmir, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Human VWF/FVIII Concentrate
Started | 41 (in this study 41 patients were screened but only 30 patients completed the study.)
Completed | 30
Not Completed | 11
Not completed — Withdrawal by Subject | 1
Not completed — Screen failure | 9
Not completed — Study termination | 1

BASELINE CHARACTERISTICS:
Arm/Group | Human VWF/FVIII Concentrate
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (18.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 7
  Poland | 2
  Oman | 2
  Romania | 8
  Turkey | 1
  Bulgaria | 1
  South Africa | 2
  Italy | 5
  India | 13

OUTCOME MEASURES:

1. Primary Outcome: Overall Hemostatic Efficacy (Success or Failure) of Wilate, Based on the Intra-operative Assessment of the Surgeon and the Post-operative Assessment by the Investigator Using a 4-point Ordinal Efficacy Scale.
Description: Efficacy of Wilate in surgical procedures was assessed intra-operatively by the surgeon and post-operatively by the investigator. The IDMC additionally conducted an independent adjudication of all hemostatic efficacy results ('secondary adjudication') and adjudicated the surgeons'/investigators' assessments of the intra- and post-operative assessments where there were discrepancies between the two assessments ('primary adjudication'). It was specified in the SAP that the study will be terminated early and success claimed if the two-sided 98.75% confidence interval (CI) for the overall success rate excludes and is greater than 0.60 (equivalent to 25 or more successes out of the 30 procedures).
Time Frame: 30 Days
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Minor Surgery: human VWF/FVIII concentrate: intravenous infusion. Dose based on subject's individual invivo-recovery
Arm/Group | Minor Surgery | Major Surgery | All Surgeries
Number analyzed (Participants) | 9 | 21 | 30
participants | 9 [NA to NA] — In this study a CI of 98.75% was used. CI: 0.569, 1.000. The success rate is 100% | 20 [NA to NA] — In this study a CI of 98.75% was used. CI: 0.704, 1.000. The success rate is 95.2% | 29 [NA to NA] — In this study a CI of 98.75% was used. CI: 0.784, 1.000. The success rate is96.7%

2. Secondary Outcome: Assessment of Intra-operative Hemostatic Efficacy
Description: The efficacy of Wilate during surgical procedures was assessed by a 4-point ordinal efficacy scale by the surgeon at the end of the surgical procedure and took the predicted versus actual blood loss and transfusion requirements into consideration. Outcome measure 1 takes the results of outcome measure 2 and 3 into consideration and is an overall assessment covering intra- and post-operative efficacy.
Time Frame: 1 Day
Measure: Number; unit: participants
Arm/Group | Intra-operative Assessment by IDMC
Number analyzed (Participants) | 30
participants | 27

3. Secondary Outcome: Post-operative Efficacy Assessment
Description: Post-operative efficacy was assessed by the investigator, covering the time period from the end of the procedure up to 24 hours following the last infusion of study medication. This assessment took the post-operative bleeding and oozing into consideration
Time Frame: up to 30 days
Measure: Number; unit: participants
Arm/Group | Post-operative Assessment by IDMC
Number analyzed (Participants) | 30
participants | 27

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each patient over a period of 1 to approximately 6 month from signing the informed consent to study completion.
Arm/Group | Human VWF/FVIII Concentrate
Serious Adverse Events (participants affected / at risk) | 2/41
Other Adverse Events (participants affected / at risk) | 29/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human VWF/FVIII Concentrate (N=41)
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human VWF/FVIII Concentrate (N=41)
Procedural Pain (Injury, poisoning and procedural complications) | 8 (10)
Nausea (Gastrointestinal disorders) | 6 (7)
Vomiting (Gastrointestinal disorders) | 6 (6)
Pain (General disorders) | 4 (4)
Pyrexia (General disorders) | 4 (4)
Hemoglobin decreased (Investigations) | 4 (6)
Hypertension (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Octapharma agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Octapharma supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial. Octapharma also reserves the right to review data prior to publishing and provide comments/changes within a certain time period.